CLINICAL TRIAL: NCT00826150
Title: Phase 1/2a, Dose-Escalation, Safety, Pharmacokinetic, and Preliminary Efficacy Study of Intraperitoneal Administration of DTA-H19 in Subjects With Advanced Stage Ovarian Cancer
Brief Title: Phase 1/2a Study of DTA-H19 in Advanced Stage Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anchiano Therapeutics Israel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-08-01
Record Dates: First submitted 2009-01-18; First posted 2009-01-21 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-05

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; H19 gene; plasmid; inodiftagene vixteplasmid
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BC-819 (Experimental): BC-819 60, 120 and 240 mg IP administration
  Interventions: Biological: BC-819

INTERVENTIONS:
Biological: BC-819 — Cohort #1: 60 mg IP weekly for 3 weeks, one week rest, then repeat for 2 more courses / 60 mg IP weekly for 3 weeks, four week rest, then repeat for 1 more course.
  Cohort #2: 120 mg IP weekly for 3 weeks, four week rest, then repeat for 1 more course.
  Cohort #3: 240 mg IP weekly for 3 weeks, four week rest, then repeat for 1 more course.
  Other Names: DTA-H19

SUMMARY:
This study is designed to assess the safety, tolerability, pharmacokinetics (PK) and preliminary efficacy of DTA-H19 administered intraperitoneally (IP) in subjects with advanced stage ovarian cancer, or primary peritoneal carcinoma

DETAILED DESCRIPTION:
This is a Phase 1/2a, open label, dose escalation, repeat dose study in 11 subjects with recurrent, platinum resistant advanced stage ovarian cancer or primary peritoneal carcinoma designed to determine the tolerability, safety, quality of life, PK, and preliminary efficacy of DTA-H19 administered intraperitoneally(IP).

Primary Objective: The primary objectives of this study are:

* To determine the maximum tolerated dose (MTD) of IP DTA-H19; and,
* To identify any dose limiting toxicities (DLTs).

Secondary Objectives: Secondary objectives of this study are:

* To determine quality of life of subjects with advanced ovarian cancer, primary peritoneal carcinoma treated with IP DTA-H19;
* To determine the the reduction in malignant ascites as measured by Ultrasound and change in frequency of parecenteses necessary.
* To determine the overall survival distribution.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and be at least 18 years of age.
* Have histopathologically documented epithelial ovarian carcinoma or primary peritoneal carcinoma with evidence of ascites.
* Have either a) platinum-refractory disease (i.e. persistent disease following completion of platinum-based primary chemotherapy) and have failed at least primary platinum-based chemotherapy; or b) platinum-resistant recurrent disease and have failed at least one regimen of second line chemotherapy.
* Be able to tolerate placement of IP catheter.
* Be at least 2 weeks from last treatment to allow recovery from prior toxicity but in the judgment of the investigator with sufficient time to ensure that the effects of prior treatments will not confound safety evaluations.
* Have a Karnofsky performance status score of ≥ 70%.
* Not be of child-bearing potential.
* Have a life expectancy of ≥ 3 months.
* Have serum creatinine < 2.0 mg/dL, total bilirubin less than the institution's 3x upper limit of normal (ULN); AST and ALT <= 2.5 x ULN,total albumin ≥ 2.5 g/dL, PT, PTT, and PT/INR within normal limits, absolute neutrophil count (ANC) > 1,500 x 103 cells/mL, platelets ≥ 100,000/mL, and hemoglobin ≥ 10 mg/dL.
* Have a biopsy specimen or an ascites fluid that is positive for H19 expression.
* Have screening procedures completed within 6-weeks before starting treatment.
* No significant history of cardiac disease, i.e., uncontrolled hypertension, unstable angina or congestive heart failure.
* - No plans to receive concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy or any other type of therapy for treatment of cancer while on this protocol.

Exclusion Criteria:

* Have evidence of extra abdominal disease with the exception of isolated small nodules (e.g., liver or pulmonary nodules) that are not causing symptoms.
* Have known brain metastases.
* Have known HIV infection.
* Have known active viral or bacterial infections.
* Have presence of any psychological, familiar, sociological, or geographical condition potentially hampering compliance with the study protocol or follow up schedule.
* Have a medical condition contraindicated for laparotomy, laparoscopy, or surgery.
* Have significant bowel involvement denoted by persistent grade 3 vomiting (≥6 episodes in 24 hrs; IV fluids, or total parenteral nutrition (TPN) indicated ≥24 hrs) after removal of ascites, inability to tolerate oral diet or medications, requirement for total parenteral nutrition, or recent (past six weeks) episode of bowel obstruction.
* Have a history of coagulopathy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tally Levy, M.D., Principal Investigator — The Edith Wolfson Medical Center; David Edelman, MD, Principal Investigator — Hadassah University Hospital; Ami Fishman, MD, Principal Investigator — Meir Medical Center; Eitan Rami, MD., Principal Investigator — Rabin Medical Center; Ofer Lavie, M.D., Principal Investigator — Carmel Medical Center; Ronnie Shapira-Frommer, MD, Principal Investigator — Sheba Medical Center
Locations (4):
- Israel (4):
  - The Edith Wolfson Medical Center, Holon
  - Hadassah University Hospital, Jerusalem
  - Meir Hospital, Kfar Saba
  - Sheba Medical Center, Tel Litwinsky

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical sites
Groups:
- BC-819 60 mg IP: 60 mg IP weekly for 3 weeks, one week rest, then repeat for 2 more courses/ 60 mg IP weekly for 3 weeks, four week rest, then repeat for 1 more course.
- BC-819 120 mg IP: 120 mg IP weekly for 3 weeks, four week rest, then repeat for 1 more course.
- BC-819 240 mg IP: 240 mg IP weekly for 3 weeks, four week rest, then repeat for 1 more course.
Period: Overall Study
Arm/Group | BC-819 60 mg IP | BC-819 120 mg IP | BC-819 240 mg IP
Started | 8 | 3 | 3
Completed | 2 | 1 | 0
Not Completed | 6 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- BC-819 60 mp IP: 60 mg IP weekly for 3 weeks, one week rest, then repeat for 2 more courses / 60 mg IP weekly for 3 weeks, four week rest, then repeat for 1 more course.
- Total: Total of all reporting groups
Arm/Group | BC-819 60 mp IP | BC-819 120 mg IP | BC-819 240 mg IP | Total
Number analyzed (Participants) | 8 | 3 | 3 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 3 | 11
  >=65 years | 3 | 0 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (12) | 61.3 (3.1) | 54.3 (7.6) | 59.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 3 | 14
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 8 | 3 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities
Description: A dose limiting toxicity (DLT) was defined as any grade 3 or greater non-hematologic AE by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE). If one subject in a cohort experienced a DLT, then three additional subjects had to be enrolled to that cohort unless a second subject in that cohort experiences a DLT. The next lower dose was to be considered the MTD.
Time Frame: 8 weeks
Population: Per Protocol data set (PP): 11 subjects who met the study inclusion and exclusion criteria, received at least one course of treatment of the investigational product and had a follow-up disease assessment comprised the PP set (5 subjects from the 60 mg cohort, 3 subjects from the 120 mg cohort; 3 subjects from the 240 mg cohort).
Measure: Count of Participants; unit: Participants
Groups:
- BC-819 60 mg IP: 60 mg IP weekly for 3 weeks, one week rest, then repeat for 2 more courses / 60 mg IP weekly for 3 weeks, four week rest, then repeat for 1 more course.
Arm/Group | BC-819 60 mg IP | BC-819 120 mg IP | BC-819 240 mg IP
Number analyzed (Participants) | 8 | 3 | 3
Participants | 0 | 0 | 0

2. Secondary Outcome: Overall Survival in ITT Population
Description: Overall survival, defined as the time from the start of treatment until the subject died, was estimated by Kaplan Meier curves.
Time Frame: 17.5 months
Population: Intent to Treat (ITT) data set: subjects who participated in the study were included in the safety and in the ITT analysis. All 14 subjects who participated in the study were included in the ITT.
Measure: Median (Full Range); unit: Months
Arm/Group | BC-819 60 mp IP | BC-819 120 mg IP | BC-819 240 mg IP
Number analyzed (Participants) | 8 | 3 | 3
Months | 3.2 [1.6 to 16.7] | 5.3 [3.2 to 8.3] | 6.5 [1.6 to 16.7]

3. Secondary Outcome: Solid Tumor Response
Description: If measurable disease was present, then the response of each marker lesion was evaluated separately and rated for response according to RECIST criteria for solid tumors.
  Complete Response: Disappearance of the target lesion. Partial Response: At least a 30% decrease in the longest diameter of the target lesion.
  Stable Disease: No sufficient shrinkage to qualify for partial response, or sufficient increase to qualify for progressive disease.
  Progressive Disease: At least a 20% increase in the longest diameter of the target lesion.
Time Frame: 6 weeks
Population: Intent To Treat (ITT) data set: subjects who participated in the study were included in the safety and in the ITT analysis. All 14 subjects who participated in the study were included in the ITT. 13 patients of the ITT population (n=14) were evaluated (one patient was not assessed for solid tumor response in the BC-819 60 mg IP Arm).
Measure: Count of Participants; unit: Participants
Arm/Group | BC-819 60 mg IP | BC-819 120 mg IP | BC-819 240 mg IP
Number analyzed (Participants) | 7 | 3 | 3
Participants
  Stable Disease | 2 | 2 | 0
  Progressive Disease | 2 | 1 | 3
  Not evaluable | 3 | 0 | 0

4. Secondary Outcome: Systemic BC-819 Pharmacokinetics (PK) by Treatment - T1/2 (Hours)
Description: Blood was collected at the indicated time points, then analyzed with a quantitative polymerase chain reaction (Q-PCR) method to quantitate the amount of plasmid present.
Time Frame: Before the start of the infusion of BC-819 and 2, 4, 6, 8, 24, and 48 hours after the start of the infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BC-819 60 mg IP | BC-819 120 mg IP | BC-819 240 mg IP
Number analyzed (Participants) | 8 | 3 | 3
hours | 12.41 (5.24) | 21.98 (12.71) | 42.04 (58.52)

5. Secondary Outcome: Systemic BC-819 Pharmacokinetics (PK) - Maximum Observed Plasma Concentration (Cmax)
Description: as for outcome 4
Time Frame: Before the start of the infusion of BC-819 and 2, 4, 6, 8, 24, and 48 hours after the start of the infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: copies/μL
Arm/Group | BC-819 60 mg IP | BC-819 120 mg IP | BC-819 240 mg IP
Number analyzed (Participants) | 8 | 3 | 3
copies/μL | 830000 (640000) | 750000 (1050000) | 430000 (340000)

6. Secondary Outcome: Systemic BC-819 Pharmacokinetics (PK) by Treatment - Tmax (Hours)
Description: as for outcome 4
Time Frame: Before the start of the infusion of BC-819 and 2, 4, 6, 8, 24, and 48 hours after the start of the infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BC-819 60 mg IP | BC-819 120 mg IP | BC-819 240 mg IP
Number analyzed (Participants) | 8 | 3 | 3
hours | 6.00 (2.14) | 2.67 (1.16) | 9.33 (12.70)

7. Secondary Outcome: Systemic BC-819 Pharmacokinetics (PK) by Treatment - AUClast
Description: as for outcome 4
Time Frame: Before the start of the infusion of BC-819 and 2, 4, 6, 8, 24, and 48 hours after the start of the infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: copies*hr/μl
Arm/Group | BC-819 60 mg IP | BC-819 120 mg IP | BC-819 240 mg IP
Number analyzed (Participants) | 8 | 3 | 3
copies*hr/μl | 1600000 (1700000) | 10600000 (15100000) | 5300000 (1900000)

8. Secondary Outcome: Systemic BC-819 Pharmacokinetics (PK) by Treatment - AUCinf
Description: as for outcome 4
Time Frame: Before the start of the infusion of BC-819 and 2, 4, 6, 8, 24, and 48 hours after the start of the infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: copies*hr/μl
Arm/Group | BC-819 60 mg IP | BC-819 120 mg IP | BC-819 240 mg IP
Number analyzed (Participants) | 8 | 3 | 3
copies*hr/μl | 1900000 (1900000) | 16200000 (24400000) | 12500000 (9800000)

9. Secondary Outcome: Overall Survival in PP
Description: as for outcome 2
Time Frame: 17.5 months
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | BC-819 60 mg IP | BC-819 120 mg IP | BC-819 240 mg IP
Number analyzed (Participants) | 5 | 3 | 3
months | 3.9 [3.1 to 16.7] | 5.3 [3.2 to 8.3] | 6.5 [4.5 to 7.4]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed over a 16 week period, starting with each participant's first treatment with IP.
Groups:
- BC-819 240 mg IP: 120 mg IP weekly for 3 weeks, four week rest, then repeat for 1 more course.
Arm/Group | BC-819 60 mg IP | BC-819 120 mg IP | BC-819 240 mg IP
All-Cause Mortality (participants affected / at risk) | 3/8 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 6/8 | 1/3 | 0/3
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BC-819 60 mg IP (N=8) | BC-819 120 mg IP (N=3) | BC-819 240 mg IP (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Elevated liver enzymes (Investigations) | 1 (1) | 0 (0) | 0 (0)
Clinical deterioration (General disorders) | 3 (3) | 0 (0) | 0 (0)
Recurrent urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Weakness and shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infection of port (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chest pain and dyspnea (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BC-819 60 mg IP (N=8) | BC-819 120 mg IP (N=3) | BC-819 240 mg IP (N=3)
Cardiac disorder (Cardiac disorders) | 1 | 2 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 6 | 2 | 1 — All other Gastrointestinal disorders excluding constipation, diarrhea, Dyspepsia, and vomiting.
General disorders and administration site conditions (General disorders) | 5 | 3 | 2 — All other general disorders and administration site conditions excluding Asthenia and general physical health deterioration.
Infections (Infections and infestations) | 1 | 1 | 0
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 3 | 0 | 0 — All other Injury, poisoning and procedural complications excluding fall
Investigations (Investigations) | 8 | 3 | 3 — All other investigations excluding those listed in this table.
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hedache (Nervous system disorders) | 2 | 0 | 1
Renal and urinary disorders (Renal and urinary disorders) | 4 | 0 | 1 — All other renal and urinary disorders excluding urinary tract infection.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 1 | 0
Asthenia (General disorders) | 4 | 2 | 0
General physical health deterioration (General disorders) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 3 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Vascular disorders (Vascular disorders) | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 4 | 1 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 0
Blood albumin decreased (Investigations) | 2 | 2 | 1
Blood calcium decreased (Investigations) | 3 | 3 | 1
Blood potassium increased (Investigations) | 3 | 1 | 0
Haemoglobin decreased (Investigations) | 3 | 0 | 1
International normalised ratio increased (Investigations) | 2 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No